CLINICAL TRIAL: NCT04222088
Title: Efficacy and Safety of Artemether-lumefantrine for the Treatment of Uncomplicated Plasmodium Falciparum Malaria and Chloroquine for Plasmodium Vivax in the Philippines From 2013-2014
Brief Title: TES of Artemether-lumefantrine for Pf and Chloroquine for Pv in the Philippines From 2013-2014
Acronym: TES
Status: Completed | Type: Observational
Sponsor: Research Institute for Tropical Medicine, Philippines (Other Government)
Collaborators: World Health Organization (Other)
Responsible Party: Principal Investigator, Fe Espino, Principal Investigator, Head of Parasitology Department, Research Institute for Tropical Medicine, Philippines
Other Study IDs: 2003-25-12_2013
Record Dates: First submitted 2019-12-15; First posted 2020-01-09 (Actual); Results first posted 2023-02-23 (Actual); Last update posted 2023-07-21 (Actual); Status verified 2023-07

CONDITIONS: Malaria; Falciparum Malaria; Vivax Malaria; Malaria Recrudescence
Keywords: malaria; TES; Plasmodium falciparum; Artemether-lumefantrine; Plasmodium vivax; Chloroquine
MeSH Terms: conditions — Malaria; Malaria, Falciparum; Malaria, Vivax | interventions — Artemether, Lumefantrine Drug Combination; Chloroquine; Primaquine

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Capillary blood (malaria blood film and filter paper)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

GROUPS / COHORTS (2):
- Patients detected with Plasmodium falciparum (Artemether-lumefantrine): Patients with mono-infection of Plasmodium falciparum with 1,000-100,000 asexual forms per µl
  Interventions: Drug: Arthemeter-lumefantrine; Drug: Primaquine
- Patients detected with Plasmodium vivax (Chloroquine): Patients with mono-infection of Plasmodium falciparum with ≥ 250 per µl
  Interventions: Drug: Chloroquine; Drug: Primaquine

INTERVENTIONS:
Drug: Arthemeter-lumefantrine — Artemether-lumefantrine will be administered for 3 days according to body weight (Days 0 and 8 hours after, 1 and 2). Dosage depending on body weight or age if weight cannot be determined.
  Dosage: 1 tablet contains 20 mg artemether and 120 mg lumefantrine Dosage per weight: 1 tablet (5 to <16kg); 2 tablets (15 to <25kg); 3 tablets (25 to <35kg), 4 tablets for >35 kg) Dosage per age, if weight cannot be determined: 1 tablet (6 months old to 3 years old); 2 tablets (4 to 8 years old); 3 tablets (9-13 years old), 4 tablets (>13 years old)
  Other Names: Coartem
  Groups: Patients detected with Plasmodium falciparum (Artemether-lumefantrine)
Drug: Chloroquine — Chloroquine will be administered according to body weight at a total dose of 25 mg base/kg over 3 days (10 mg base/kg on Day 0; 10 mg base/kg on Day 1 and 5 mg base/kg on Day 2). Correct drug dosage will be determined using the dosing chart (in accordance with national treatment guidelines)
  Groups: Patients detected with Plasmodium vivax (Chloroquine)
Drug: Primaquine — For Pf patients, primaquine at 0.75 mg base/kg body weight single dose will be given on Day 3 for Pf patients; For Pv patients primaquine will be withheld for 28 days and will be given after Day 28 follow-up, at 0.25 mg base/kg per day for 14 days.

SUMMARY:
An antimalarial drug efficacy trial was conducted for artemether-lumefantrine (AL) and chloroquine (CQ) in the three (3) municipalities (Bataraza, Brookes and Rizal) of Palawan. Study subjects are febrile individuals between > 6 months old and 59 years old with confirmed uncomplicated P. falciparum or P. vivax infections. Patients with P. falciparum was treated with Artemether-lumefantrine administered 3 days (Days 0, 1 and 2) according to body weight. Primaquine at 0.75 mg base/kg body weight single dose was given on Day 3. For Plasmodium vivax patients chloroquine were administered according to body weight at a total dose of 25 mg/kg over 3 days (10 mg/kg on Day 0; 10 mg/kg on Day 1 and 5 mg/kg on Day 2), and primaquine following the National Treatment Guidelines.

During the period that this report covers, 84 and 75 patients met the inclusion criteria for Pf and Pv respectively. Clinical and parasitological parameters were monitored over a 28-day follow-up period for both drugs.

The presence of only 1 Late Clinical Failure (LCF) of P. falciparum parasitemia out of 84 enrolled patients and 2 Late Parasitological Failure (LPF) of P. vivax patients out of 75 enrolled patients within the 28 days follow up suggest that both drugs are still efficacious.

DETAILED DESCRIPTION:
In 2002, the Philippines changed its antimalarial drug policy to the combination treatment, CQ+SP as 1st-line treatment and artemether-lumefantrine as 2nd-line treatment. The DOH prescribed the use of artemether-lumefantrine (AL) combination as the second-line drug, limiting its use only in the treatment of confirmed Plasmodium falciparum until a further study on its efficacy was done before making it as the first-line treatment. Consequently, AL became the first-line drug for falciparum malaria in the 2009 revised drug policy. The DOH in the past 6 years (2002-2007) adopted the use of AL in the highly endemic areas of the country and conducted therapeutic efficacy studies (TES) in 3 sentinel sites: Kalinga-Isabela, Palawan, and several Mindanao provinces showing 97-100% efficacy. Whereas CQ+SP showed variability and declining efficacy, results ranged from 70%-95% (CARAGA region). In Sultan Kudarat province, results in 2006-2007 showed 90% efficacy of CQ+SP and 96% for AL for falciparum malaria.

In the 2009 drug policy, chloroquine (CQ) remains the primary treatment for P. vivax malaria, with primaquine as an anti-relapse drug. Previous studies (1999-2005) elsewhere in the country have shown 100% efficacy of CQ or the CQ+PQ combination. However, in 2011, recurrence of parasitemia was observed in one of 117 enrolled patients in Palawan. The last TES of AL as a first-line drug of choice for falciparum malaria was made in 2007. This study will update this drug's efficacy for this parasite and that of P. vivax.

STUDY OBJECTIVES The general objective of this study is to assess the therapeutic efficacy and safety artemether-lumefantrine for the treatment of uncomplicated P. falciparum infections and of chloroquine for the treatment of P. vivax infections in Palawan province, the Philippines from 2013-2014.

The specific objectives are:

* To measure the clinical and parasitological efficacy of artemether-lumefantrine (AL) among patients aged between > 6 months and 59 years old suffering from uncomplicated falciparum malaria, by determining the proportion of patients with Early Treatment Failure (ETF), Late Clinical Failure (LTF), Late Parasitological Failure (LPF), or with an Adequate Clinical and Parasitological Response (ACPR) as indicators of efficacy;
* To measure the clinical and parasitological efficacy of Chloroquine among patients aged between > 6 months and 59 years old suffering from vivax malaria, by determining the proportion of patients with clinical and parasitological failure, or with an Adequate Clinical and Parasitological Response (ACPR) as indicators of efficacy;
* To evaluate the incidence of adverse events;
* To formulate recommendations to enable the Department of Health to make informed decisions about the possible need for updating of the current national antimalarial treatment guidelines.

STUDY DESIGN The design of this surveillance study is a one-arm, prospective evaluation of the clinical and parasitological response to directly observed treatment for uncomplicated falciparum and vivax malaria. Individuals with uncomplicated malaria who meet the study inclusion criteria will be enrolled, treated on-site with AL, and monitored for a period of 28 days if they have falciparum malaria, and with chloroquine if with vivax malaria, and monitored for a period of 28 days. The follow-up consists of a fixed schedule of check-up visits and corresponding clinical and laboratory examinations. Study patients have been classified as therapeutic failures (early or late) or adequate responders based on the results of these assessments. The proportion of patients experiencing a therapeutic failure during the follow-up period has been used to estimate the efficacy of the study drug(s). Polymerase Chain Reaction (PCR) analysis will also help distinguish between a true recrudescence due to treatment failure and episodes of re-infection.

STUDY AREA The study was conducted in the Rural Health Units (RHU) of Bataraza, Brookes Point, and Rio Tuba Nickel Foundation Inc. Hospital (RTNFI). However, due to the difficulty of recruiting patients in RTNFI, recruitment was stopped in October 2013 and was replaced by the RHU of Rizal. Several factors influenced the selection of sites: adequate numbers of patients with symptomatic, uncomplicated P. falciparum or P. vivax malaria; willingness and availability of the selected health care facility staff to participate in the trial and to support the work with laboratory space; access of patients to the health facility for weekly follow-ups; availability of the Municipality Health Officer (MHO), the nurse and a trained Medical Technologist to take responsibility for conducting the trail, and security.

SAMPLE SIZE Treatment failure to AL in the area being 0-5 %, 5% has been chosen as the estimated therapeutic failure rate of the drug. At a confidence level of 95% and with precision around the estimate of 10%, 18 patients will be needed. With a 20% increase to allow losses to follow-up and withdrawals during the 28-day follow-up period, 22 patients need to be included. But in order for the sample to be representative, a minimum of 50 P. falciparum and 50 P. vivax patients need to be included and a maximum of 75 patients for Plasmodium falciparum and 75 Plasmodium vivax will be enrolled.

SAMPLING TECHNIQUE All individuals who consulted at the selected rural health units met the inclusion criteria and had none of the exclusion criteria were included in the study.

DATA MANAGEMENT The principal investigator has ensured that the study protocol is strictly adhered to throughout and that all data are collected and recorded correctly on the CRF. Laboratory and clinical data have been recorded on a daily basis in the CRF designed for the study. Data that are derived from source documents are consistent with the source documents or the discrepancies were explained. Any changes or corrections to a CRF were dated and explained and did not obscure the original entry. All CRF was checked for completeness. After the study was completed, data were entered onto a database using double independent data entry. The data were stored in a computer database maintaining confidentiality in accordance with the national data legislation.

ETHICAL CONSIDERATIONS Participants were recruited after the study received favorable approval of the protocol, participant information sheet, and written informed consent form from RITM Institutional Review Board (IRB). The study document versions given written approval by the IRB were used. The study was carried out according to the ethical guidelines in the Declaration of Helsinki (version 2008), applicable guidelines of ICH-GCP (E6); and applicable regulations of the Department of Health, Manila. The participant's written informed consent was secured before enrolment and prior to initiating procedures specific to this study. For potential participants below 18 years old, this consent was obtained from either parent or a legally accepted guardian. An independent witness was present during the process of obtaining informed consent from a participant or parents/legal guardian who was illiterate.

ELIGIBILITY:
Inclusion Criteria:

* Above 6 months old to 59 years old;
* Mono-infection with P. falciparum (1000-100 000 asexual forms per µl) and P. vivax (≥250/ul)
* Axillary temperature ≥37.5 °C or oral/rectal temperature of ≥38 °C;
* Glucose-6-dehydrogenase (G6PD) test normal for vivax patients if available
* Ability to swallow medication;
* Ability and willingness to comply with the study protocol for the duration of the study and to comply with the study visit schedule;
* Informed consent from the patient or from a parent or legal guardian in the case of children less than 18 years old;
* Informed assent from any minor participant aged 12 - 17 years; and
* Consent for pregnancy testing from female of child-bearing potential and from their parent or guardian if under 18 years old.

Exclusion Criteria:

* Presence of general danger signs among children <5 years old or other signs of severe and complicated falciparum malaria according to current WHO definitions
* Mixed Plasmodium species;
* Presence of severe malnutrition
* Presence of febrile conditions due to diseases other than malaria (measles, acute lower tract respiratory infection, severe diarrhea with dehydration, etc.), or other known underlying chronic or severe diseases (e.g. cardiac, renal, hepatic diseases, HIV/AIDS)
* History of hypersensitivity reactions to any of the drug(s) being tested or used as alternative treatment.

Ages: 6 Months to 59 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: The population of interest consists of patients aged between > 6 months to 59 years old diagnosed with uncomplicated falciparum and vivax malaria attending the study health clinic, and having given, or whose parents or legal guardians have given an informed consent for study inclusion and assent in children as appropriate.
Sampling Method: Non-Probability Sample
Enrollment: 159 (Actual)
Dates: Start 2013-05-01 (Actual); Primary Completion 2014-12-30 (Actual); Study Completion 2014-12-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Fe Esperanza Caridad J Espino, MD, PhD, Principal Investigator — Research Institute for Tropical Medicine, Philippines

IPD SHARING:
Plan to Share IPD: Yes
The IPD will be shared with Data Transfer Agreement and IRB Approval
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Data information will be provided upon request
Access Criteria: Data Transfer

REFERENCES:
- [Background] Council for International Organizations of Medical Sciences. International ethical guidelines for biomedical research involving human subjects. Bull Med Ethics. 2002 Oct;(182):17-23. PMID 14983848
- [Background] World Medical Association. World Medical Association Declaration of Helsinki: ethical principles for medical research involving human subjects. JAMA. 2013 Nov 27;310(20):2191-4. doi: 10.1001/jama.2013.281053. No abstract available. PMID 24141714

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study Sites:
  1. Rural Health Unit, Bataraza, Palawan
  2. Rural Health Unit, Rizal, Palawan
  3. Rural Health Unit, Brooke's Point Palawan
  Study Period: May 2013 - December 2014
Pre-assignment Details: The number of total patients enrolled/started (159) is different from the total number of patients who completed the study (149) due to lost to follow-up and withdrawal of the patients in the middle of the study. Thus, all 159 patients have baseline characteristics and adverse effects, but only 149 patients who completed the study have outcome measurements.
Groups:
- Artemether-lumefantrine (Coartem™) + Primaquine: Administered to patients with mono-infection of Plasmodium falciparum with 1000-100 000 asexual forms per µl. Coartem™: 20/120 mg per tablet was administered 3 days (Days 0, 1 and 2) according to body weight. For patients with weight of 5 to <15kg, 15 to <25kg, 25 to <35kg, or ≥35kg, tablets of 1, 2, 3, or 4 will be given respectively. At day 3, primaquine at 0.75 mg base/kg body weight single dose will be given .
- Chloroquine + Primaquine: Administered to patients with mono-infection of Plasmodium vivax with parasite count of ≥ 250 per µl, Chloroquine 150 mg base tablet was administered according to body weight at a total dose of 25 mg/kg over 3 days (10 mg/kg on Day 0; 10 mg/kg on Day 1 and 5 mg/kg on Day 2). After 28 days of follow-up, primaquine will be given for 14 days.
Period: Overall Study
Arm/Group | Artemether-lumefantrine (Coartem™) + Primaquine | Chloroquine + Primaquine
Started | 84 | 75
Completed | 75 | 74
Not Completed | 9 | 1
Not completed — Lost to Follow-up | 5 | 1
Not completed — Withdrawal by Subject | 4 | 0

BASELINE CHARACTERISTICS:
Groups:
- Artemether-lumefantrine (Coartem™) + Primaquine: Administered to patients with mono-infection of Plasmodium falciparum with 1000-100 000 asexual forms per µl. Coartem™: 20/120 mg per tablet was administered 3 days (Days 0, 1 and 2) according to body weight. For patients with weight of 5 to <15kg, 15 to <25kg, 25 to <35kg, or ≥35kg, tablets of 1, 2, 3, or 4 will be given respectively. At day 3, primaquine at 0.75 mg base/kg body weight single dose will be given.
- Total: Total of all reporting groups
Arm/Group | Artemether-lumefantrine (Coartem™) + Primaquine | Chloroquine + Primaquine | Total
Number analyzed (Participants) | 84 | 75 | 159
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: Analysis of population was categorically subdivided depending on the period of enrollment
  years | 13.52 (12.25) | 10.26 (9.66) | 11.98 (11.19)
Age, Continuous [Mean (Full Range); unit: years] — Population: Analysis of population was categorically subdivided depending on the period of enrollment
  years | 13.52 [1 to 53] | 10.26 [0 to 42] | 11.98 [0 to 53]
Age, Customized [Count of Participants; unit: Participants] — Population: Analysis of population was categorically subdivided depending on the period of enrollment
  Participants
    >15 years old | 20 | 22 | 42
    5 - 15 years old | 48 | 24 | 72
    <5 years old | 16 | 29 | 45
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Analysis of population was categorically subdivided depending on the period of enrollment
  Participants
    Female | 37 | 21 | 58
    Male | 47 | 54 | 101
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Weight (mean, sd) [Mean (Standard Deviation); unit: kg] — Population: Analysis of population was categorically subdivided depending on the period of enrollment
  kg | 27.23 (15.62) | 25.58 (17.72) | 26.45 (16.61)
Weight (mean, full range) [Mean (Full Range); unit: kg] — Population: Analysis of population was categorically subdivided depending on the period of enrollment
  kg | 27.23 [7.8 to 78] | 25.58 [5 to 62.7] | 26.45 [5 to 78]
Temperature Day 0(mean, SD) [Mean (Standard Deviation); unit: degrees celcius] — Population: Analysis of population was categorically subdivided depending on the period of enrollment
  degrees celcius | 38.1 (1.3) | 38.0 (1.1) | 38.0 (1.2)
Temperature Day 0 (mean, full range) [Mean (Full Range); unit: degrees Celcius] — Population: Analysis of population was categorically subdivided depending on the period of enrollment
  degrees Celcius | 38.1 [36 to 41.2] | 38.0 [36.1 to 41.5] | 38.0 [36 to 41.5]
Parasitemia Day 0 [Geometric Mean (Full Range); unit: uL] — Population: Analysis of population was categorically subdivided depending on the period of enrollment
  uL | 16860 [1304 to 99460] | 5514 [280 to 32862] | 9952 [280 to 99460]

OUTCOME MEASURES:

1. Primary Outcome: Early Treatment Failure (ETF)
Description: The classification of treatment outcomes will be based on an assessment of the parasitological and clinical outcomes of antimalarial treatment according to the latest guidelines of WHO. Accordingly, all patients will be classified as having an Early Treatment Failure by microscopy results P without PCR correction
  * Development of danger signs or severe malaria on day 1, day 2, or day 3 in the presence of parasitemia;
  * Parasitaemia on day 2 higher than day 0 count irrespective of axillary temperature;
  * Parasitaemia on day 3 with axillary temperature ≥37.5 ºC;
  * Parasitaemia on day 3 ≥25% of count on day 0.
Time Frame: Day 1-3
Population: Analysis of population is categorically subdivided depending on the period of enrollment of participants to the study
Measure: Number (95% Confidence Interval); unit: participants
Arm/Group | Artemether-lumefantrine (Coartem™) + Primaquine | Chloroquine + Primaquine
Number analyzed (Participants) | 75 | 74
participants | 0 [0 to 4.8] | 0 [0 to 4.9]

2. Primary Outcome: Late Clinical Failure (LCF)
Description: Patients with late clinical failure without PCR correction:
  * Development of danger signs or severe malaria on any day from day 4 to day 28 in the presence of parasitaemia, without previously meeting any of the criteria of Early Treatment Failure;
  * Presence of parasitemia and axillary temperature ≥37.5 ºC (or history of fever in low/moderate transmission areas) on any day from day 4 to day 28, without previously meeting any of the criteria of Early Treatment Failure.
Time Frame: Day 4-28
Population: Analysis of population is categorically subdivided depending on the period of enrollment of participants in the study
Measure: Number (95% Confidence Interval); unit: participants
Arm/Group | Artemether-lumefantrine (Coartem™) + Primaquine | Chloroquine + Primaquine
Number analyzed (Participants) | 75 | 74
participants | 1 [0 to 7.2] | 0 [0 to 4.9]

3. Primary Outcome: Late Parasitological Failure (LPF)
Description: Patients with late parasitological failure without PCR correction:
  • Presence of parasitemia on any day from day 7 to day 28 and axillary temperature <37.5 ºC, without previously meeting any of the criteria of Early Treatment Failure or Late Clinical Failure.
Time Frame: day 7 to day 28
Population: Analysis of population is categorically subdivided depending on the period of enrollment of participants in the study
Measure: Number (95% Confidence Interval); unit: participants
Arm/Group | Artemether-lumefantrine (Coartem™) + Primaquine | Chloroquine + Primaquine
Number analyzed (Participants) | 75 | 74
participants | 0 [0 to 4.8] | 2 [0.3 to 9.4]

4. Primary Outcome: Adequate Clinical and Parasitological Response (ACPR)
Description: Adequate Clinical and Parasitological Response (ACPR): Absence of parasitemia on day 28 irrespective of axillary temperature without previously meeting any of the criteria of Early Treatment Failure or Late Clinical Failure or Late Parasitological Failure.
Time Frame: Day 0-28
Population: Analysis of population is categorically subdivided depending on the period pf enrollment of the participant in the study
Measure: Count of Participants; unit: Participants
Arm/Group | Artemether-lumefantrine (Coartem™) + Primaquine | Chloroquine + Primaquine
Number analyzed (Participants) | 75 | 74
Participants | 74 | 72

ADVERSE EVENTS:
Time Frame: Study patients will be observed for 30 minutes after drug administration for adverse reactions or vomiting. The study patient will be monitored during the whole duration of the study: 28 days for patients with Pf infections and 42 days for patients with Pv infections.
Description: Information concerning the adverse event and symptomatic treatment given must be recorded on the case record form (CRF). If the adverse event is serious, the principal investigator must notify the sponsor or its designee immediately and the reporting procedures described in the safety section must be followed.
Arm/Group | Artemether-lumefantrine (Coartem™) + Primaquine | Chloroquine + Primaquine
All-Cause Mortality (participants affected / at risk) | 0/84 | 0/75
Serious Adverse Events (participants affected / at risk) | 0/84 | 0/75
Other Adverse Events (participants affected / at risk) | 0/84 | 0/75

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-07-19): https://cdn.clinicaltrials.gov/large-docs/88/NCT04222088/Prot_SAP_000.pdf